CLINICAL TRIAL: NCT06208332
Title: Photo-Narrative Pilot Randomized Controlled Trial
Brief Title: Photo-Narrative Study
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00004439
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Child Development Disorder; Critical Illness; Neurologic Disorder
Keywords: pediatric palliative care; communication; severe neurological impairment
MeSH Terms: conditions — Developmental Disabilities; Critical Illness; Nervous System Diseases; Communication; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photo-Narrative (Experimental)
  Interventions: Behavioral: Photo-Narrative
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Photo-Narrative — Photo-Narratives include 1-3 photos of the pediatric patient and their family to tell a story about palliative care topics that are shared with the child's clinicians.
  Arms: Photo-Narrative

SUMMARY:
The objective of this study is to conduct a pilot randomized controlled trial (RCT) of a photo-narrative communication intervention developed by our study team with patients/parents of children with severe neurological impairment (SNI) and their pediatric intensive care unit (PICU) clinicians to assess feasibility, acceptability, and early efficacy.

ELIGIBILITY:
Patients

Inclusion Criteria:

* ages 3 months-25 years
* severe neurological impairment (including congenital/chromosomal, chronic central nervous system static or progressive conditions, or child >6 months after severe traumatic brain injury
* admitted to the pediatric ICU at Seattle Children's and with medical team permission to approach
* expected length of stay >1 week
* life expectancy >4 weeks
* previous discharge home

Parents

Inclusion Criteria:

* parent/legal guardian
* English and/or Spanish speaking (most common languages spoken at SCH making up 95% of patients and families)
* >18 years of age

Clinicians

Inclusion Criteria:

* licensed physicians, fellows, residents, advanced practice nurse practitioners, nurses, or respiratory therapists
* working in the pediatric ICU at Seattle Children's Hospital

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 30 months
  Defined as >70% enrollment [enrolled parents/total approached] and completion [parents completing intervention/total randomized to the intervention].
Acceptability | 30 month
  Defined as >70% of the intervention parents likely or very likely to recommend the intervention to others/total randomized].

CONTACTS AND LOCATIONS:
Overall Officials: Jori Bogetz, MD, Principal Investigator — Seattle Children's Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allen J, Brenner M, Hauer J, Molloy E, McDonald D. Severe Neurological Impairment: A delphi consensus-based definition. Eur J Paediatr Neurol. 2020 Nov;29:81-86. doi: 10.1016/j.ejpn.2020.09.001. Epub 2020 Sep 11. PMID 32951992
- [Background] Feudtner C, Kang TI, Hexem KR, Friedrichsdorf SJ, Osenga K, Siden H, Friebert SE, Hays RM, Dussel V, Wolfe J. Pediatric palliative care patients: a prospective multicenter cohort study. Pediatrics. 2011 Jun;127(6):1094-101. doi: 10.1542/peds.2010-3225. Epub 2011 May 9. PMID 21555495
- [Background] Berry JG, Poduri A, Bonkowsky JL, Zhou J, Graham DA, Welch C, Putney H, Srivastava R. Trends in resource utilization by children with neurological impairment in the United States inpatient health care system: a repeat cross-sectional study. PLoS Med. 2012 Jan;9(1):e1001158. doi: 10.1371/journal.pmed.1001158. Epub 2012 Jan 17. PMID 22272190
- [Background] Moreau JF, Fink EL, Hartman ME, Angus DC, Bell MJ, Linde-Zwirble WT, Watson RS. Hospitalizations of children with neurologic disorders in the United States. Pediatr Crit Care Med. 2013 Oct;14(8):801-10. doi: 10.1097/PCC.0b013e31828aa71f. PMID 23842588
- [Background] DeCourcey DD, Silverman M, Oladunjoye A, Balkin EM, Wolfe J. Patterns of Care at the End of Life for Children and Young Adults with Life-Threatening Complex Chronic Conditions. J Pediatr. 2018 Feb;193:196-203.e2. doi: 10.1016/j.jpeds.2017.09.078. Epub 2017 Nov 22. PMID 29174080
- [Background] Nolan R, Luther B, Young P, Murphy NA. Differing perceptions regarding quality of life and inpatient treatment goals for children with severe disabilities. Acad Pediatr. 2014 Nov-Dec;14(6):574-80. doi: 10.1016/j.acap.2014.02.012. Epub 2014 May 6. PMID 24816425
- [Background] Bogetz JF, Trowbridge A, Lewis H, Jonas D, Hauer J, Rosenberg AR. Forming Clinician-Parent Therapeutic Alliance for Children With Severe Neurologic Impairment. Hosp Pediatr. 2022 Mar 1;12(3):282-292. doi: 10.1542/hpeds.2021-006316. PMID 35141756
- [Derived] Bogetz J, Ayala E, Anderson J, Morris L, Barton KS, Bradford MC, Zhou C, Yi-Frazier J, Watson RS, Rosenberg AR. A photo-narrative intervention protocol for clinicians and parents of children with severe neurological impairment in the PICU. Contemp Clin Trials Commun. 2025 Feb 11;44:101455. doi: 10.1016/j.conctc.2025.101455. eCollection 2025 Apr. PMID 40034723

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT06208332/Prot_SAP_000.pdf